CLINICAL TRIAL: NCT01363687
Title: The Effect of Remote Postconditioning on Graft Function in Patients Undergoing Living-related Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011-03-047
Record Dates: First submitted 2011-05-23; First posted 2011-06-01 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Transplantation; Ischemic Reperfusion Injury; Remote Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic postconditioning group (Experimental): Recipients receive remote ischemic postconditioning after declamping of renal artery during kidney transplantation
  Interventions: Device: remote ischemic postconditioning
- Control group (No Intervention): Patients who have a deflated cuff placed on the upper limb free of arteriovenous fistula during the surgery

INTERVENTIONS:
Device: remote ischemic postconditioning — Remote ischemic postconditioning consists of three 5-min cycles of upper limb ischemia, which was induced by an automated cuff-inflator placed on the upper limb free of arteriovenous fistula and inflated to 250 mm Hg, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Arms: Remote ischemic postconditioning group

SUMMARY:
The purpose of this study is to investigate whether upper limb ischemic postconditioning can improve renal function and decrease ischemic-reperfusion injury in patients undergoing living donor kidney transplantation.

DETAILED DESCRIPTION:
Ischemic reperfusion injury after kidney transplantation is a common clinical problem associated with a high morbidity and mortality. To reduce the adverse effect of ischemic reperfusion injury after organ transplantation, various strategies including ischemic preconditioning or postconditioning. Remote ischemic postconditioning is one of such strategies where brief ischemic reperfusion injury of one organ protects other organs from sustained ischemic reperfusion injury. Remote ischemic postconditioning of the limb with a tourniquet is a safe and convenient method of postconditioning organs against ischemic reperfusion injury. However, the efficacy of remote ischemic postconditioning in patients undergoing living donor kidney transplantation needs to be established. Therefore, we investigate the efficacy of remote ischemic postconditioning of the upper limb with a tourniquet in recipients of kidney transplantation by measuring the markers of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing elective living donor kidney transplantation
* subjects older than 20 yrs who can give written informed consent

Exclusion Criteria:

* re-transplant recipients
* those with peripheral vascular disease affecting the upper limbs free of arteriovenous fistula

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
renal function of recipient after living-related kidney transplantation | 1 day before surgery
  serum creatinine concentration and urine output
renal function of recipient after living-related kidney transplantation | at 2 h after declaming of renal artery
  serum creatinine concentration and urine output
renal function of recipient after living-related kidney transplantation | at 6 h after declaming of renal artery
  serum creatinine concentration and urine output
renal function of recipient after living-related kidney transplantation | at 12 h after declaming of renal artery
  serum creatinine concentration and urine output
renal function of recipient after living-related kidney transplantation | at 24 h after declaming of renal artery
  serum creatinine concentration and urine output
renal function of recipient after living-related kidney transplantation | at 48 h after declaming of renal artery
  serum creatinine concentration and urine output
renal function of recipient after living-related kidney transplantation | at 72 h after declaming of renal artery
  serum creatinine concentration and urine output

SECONDARY OUTCOMES:
Biomarkers of acute kidney injury | before surgery and at 2, 6, 12 h after declaming of renal artery
  biomarkers of acute kidney injury: Plasma cystatin-C, Urine IL-18, Urine Neutrophil gelatinase-associated lipocalin (NGAL)
Hemodynamic parameters | before surgery and at 2, 6, 12, 24, 48, 72 h after declaming of renal artery
  arterial blood pressure, heart rate, central venous pressure, pulse oximetry
outcome of kidney transplantation | at 72 h after declaming of renal artery
  number of acute rejection or number of delayed graft function
postoperative hospital stay | at postoperative day 60
  length of postoperative hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hwan Lee, M.D.,Ph.D., Study Director — Samsung Medical Center; Won Ho Kim, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Seoul Hospital, Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim WH, Lee JH, Kim GS, Sim HY, Kim SJ. The effect of remote ischemic postconditioning on graft function in patients undergoing living donor kidney transplantation. Transplantation. 2014 Sep 15;98(5):529-36. doi: 10.1097/TP.0000000000000098. PMID 24770616